CLINICAL TRIAL: NCT06626022
Title: A Phase 3, Multicenter, International, Non-inferiority, Randomized Clinical Trial Comparing Screening for Prostate Cancer Using High Resolution Micro-ultrasound Versus Multiparametric Magnetic Resonance Imaging (MUSIC-Screen)
Brief Title: Screening for Prostate Cancer Using High Resolution Micro-ultrasound Versus Multiparametric Magnetic Resonance Imaging.
Acronym: MUSIC-Screen
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: HREBA.CC-24-0325
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer Screening

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MRI (Active Comparator)
  Interventions: Device: MRI
- microUltransound (Experimental)
  Interventions: Device: ExactVu

INTERVENTIONS:
Device: MRI — Standard prostate mpMRI.
  Arms: MRI
Device: ExactVu — microUltrasound
  Arms: microUltransound

SUMMARY:
The purpose of this study is to compare whether the FDA and Health Canada approved microUS is as effective as the currently used option (MRI) for imaging the prostate gland. Participants will be randomized into two groups to compare the imaging results of the current standard of care MRI and the new microUS. The study is looking to identify the most effective imaging modality to help guide whether you progress to have a prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex;
2. Age 50-70;
3. PSA 3-20 and/or abnormal DRE;
4. Biopsy naïve.

Exclusion Criteria:

1. Prior personal history of prostate cancer;
2. Prior prostate imaging using microUS or MRI;
3. Contraindication to microUS or MRI;
4. Testosterone replacement therapy within last 12 months; or
5. Androgen deprivation therapy within last 12 months.

Ages: 50 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1284 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2029-11-30 (Estimated)

PRIMARY OUTCOMES:
Detection of Clinically significant prostate cancer. | Once enrolled, men will be followed for 1 year after the imaging test.
  The primary objective of this trial is to determine if a screening pathway using microUS is non-inferior to a pathway using MRI for the detection of clinically significant prostate cancer, defined as Gleason Grade Group 2 or more.

CONTACTS AND LOCATIONS:
Locations (4):
- University of California, Los Angeles (UCLA), Los Angeles, California, United States
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - CIUSSS du Nord-de-l'Île-de-Montréal, Montréal, Quebec

IPD SHARING:
Plan to Share IPD: No